CLINICAL TRIAL: NCT00764907
Title: A Randomized Trial of the I-BFM-SG for the Management of Childhood Non-B Acute Lymphoblastic Leukemia
Brief Title: Risk-Adjusted Combination Chemotherapy in Treating Young Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000613220; MOTOL-ALL-IC-BFM-2002; EU-20871
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia
Keywords: T-cell childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Vindesine

ARMS (3):
- Arm I (Experimental): During reinduction, patients receive 1 course of protocol II.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: thioguanine; Drug: vincristine sulfate
- Arm II (Experimental): During reinduction, patients receive 2-3 course of protocol III and interim maintenance therapy.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: thioguanine; Drug: vincristine sulfate
- Arm III (Experimental): During reinduction, patients are receive 2 courses of protocol II and interim maintenance therapy OR 3-block consolidation regimen and 1 course of protocol II.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine

INTERVENTIONS:
Drug: asparaginase — Given IV during reinduction
Drug: cyclophosphamide — Given IV during reinduction
Drug: cytarabine — Given IV during reinduction
Drug: daunorubicin hydrochloride — Given IV during reinduction
  Arms: Arm III
Drug: dexamethasone — Given IV or orally during reinduction
Drug: doxorubicin hydrochloride — Given IV during reinduction
Drug: etoposide — Given IV during reinduction
  Arms: Arm III
Drug: ifosfamide — Given IV during reinduction
  Arms: Arm III
Drug: leucovorin calcium — Given IV during reinduction
  Arms: Arm III
Drug: mercaptopurine — Given orally during reinduction
  Arms: Arm II; Arm III
Drug: methotrexate — Given orally during reinduction
Drug: prednisone — Given intrathecally during reinduction
  Arms: Arm III
Drug: thioguanine — Given orally during reinduction
Drug: vincristine sulfate — Given IV during reinduction
Drug: vindesine — Given IV during reinduction
  Arms: Arm III

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. A donor stem cell transplant may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving combination chemotherapy before the transplant helps stop the growth of cancer cells and stop the patient's immune system from rejecting the donor's stem cells. It is not yet known which combination chemotherapy regimen is more effective in treating young patients with acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is studying different risk-adjusted combination chemotherapy regimens in treating young patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test in a randomized way the type and intensity of reintensification therapy for pediatric patients with acute lymphoblastic leukemia in each risk group: standard-risk (SR), intermediate-risk (IR), and high-risk (HR) group.
* To compare two shorter elements of reintensification (protocol III x 2 courses) to one (protocol II x 1 course) in terms of effectiveness when cumulative dose of most drugs are the same in both regimen in patients in the standard-risk group.
* To determine if the increased risk of failure in patients in the intermediate-risk group can be curtailed by a third reintensification element (protocol III x 3 courses vs protocol II x 1 course).
* To determine if the three reintensification elements (protocol III x 3 courses) achieve the same or better results in high-risk group patients, as compared with current applied HR approach in Berlin-Frankfurt-Münster Group (BFM) or Italian Association of Pediatric Hematology and Oncology (AIEOP).

OUTLINE: This is a partially randomized, multicenter study. Patients are stratified according to risk group (standard risk [SR] vs intermediate risk [IR] vs high risk [HR]). Patients are randomized in reinduction part of the treatment.

* Induction therapy:

  * Protocol I' (SR B-cell precursor [BCP] ALL ): Patients receive methotrexate intrathecally (IT) on days 1, 12, and 33 (and possibly on days 18 and 27); prednisone or prednisolone orally or IV on days 1-28 followed by a taper; vincristine sulfate IV on days 1, 8, 15, 22, and 29; daunorubicin hydrochloride IV over 1 hour on days 8 and 15; and asparaginase IV over 1 hour on days 12, 15, 18, 21, 24, 27, 30, and 33. Patients then receive cyclophosphamide IV over 1 hour on days 36 and 64; oral mercaptopurine once daily on days 36-63; cytarabine IV continuously on days 38-41, 45-48, 52-55, and 59-62; and methotrexate IT on days 45 and 59.
  * Protocol I (SR T-cell ALL, IR, or HR): Patients receive therapy as in Protocol I' except that they also receive daunorubicin hydrochloride on days 22 and 29.

Approximately 2 weeks after completion of induction therapy, patients proceed to consolidation therapy.

* Consolidation: Patients who have achieved complete cytomorphologic remission proceed to protocol mM or protocol M. Patients in HR group proceed to 3-block consolidation regimen.

  * Protocol mM (BCP-ALL) (SR or IR): Patients receive oral mercaptopurine once daily on days 1-56; medium-dose methotrexate IV over 24 hours and methotrexate IT on days 8, 22, 36, and 50; and leucovorin calcium IV every 6 hours on days 9, 23, 37, and 51.
  * Protocol M (T-cell ALL) (SR or IR): Patients receive mercaptopurine, methotrexate IT, and leucovorin calcium as in protocol mM, and they also receive high-dose (HD) methotrexate IV over 24 hours on days 8, 22, 36, and 50.
  * 3-block consolidation regimen (HR): Patients receive 3 regimen blocks with 2 weeks between blocks. Treatment continues in the absence of unacceptable toxicity.

    * Block HR-1': Patients receive dexamethasone orally or IV 3 times daily on days 1-5; vincristine sulfate IV on days 1-6; HD methotrexate IV over 24 hours on day 1; leucovorin calcium IV every 6 hours, beginning 42 hours after the start of HD methotrexate, for 3 doses; cyclophosphamide IV over 1 hour, every 12 hours, on days 2-4; HD cytarabine IV over 3 hours, every 12 hours, on day 5 (2 doses); asparaginase IV over 2 hours on days 6 and 11; and triple intrathecal therapy (TIT) comprising methotrexate, cytarabine, and prednisone, 3 times on day 1.
    * Block HR-2': Patients receive dexamethasone, HD methotrexate, leucovorin calcium, and asparaginase as in block HR-1'. Patients receive TIT once on day 1 (CNS-negative patients) or twice on days 1 and 5 (CNS-positive patients). Patients also receive vindesine IV on days 1 and 6; ifosfamide IV over 1 hour, every 12 hours, on days 2-4; and daunorubicin hydrochloride IV over 24 hours on day 5.
    * Block HR-3': Patients receive dexamethasone and asparaginase as in block HR-1'; TIT 3 times on day 5; HD cytarabine IV over 3 hours, every 12 hours, on days 1 and 2; and etoposide IV over 1 hour, every 12 hours, on days 3-5.

Approximately 2 weeks after completion of consolidation therapy, patients proceed to reinduction therapy.

* Reinduction (randomized): Patients in continuous complete remission proceed to protocol II or III. Patients from SR and IR group are randomized to arms I and II; patients from HR group are randomized to arms II and III.

  * Arm I (protocol II x 1 course) (SR-1 or IR-1): Patients receive dexamethasone orally or IV on days 1-21 followed by a taper; vincristine sulfate IV and doxorubicin hydrochloride IV over 1 hour on days 8, 15, 22, and 29; asparaginase IV over 1 hour on days 8, 11, 15, and 18; and methotrexate IT on days 1 and 18. Patients then receive cyclophosphamide IV over 1 hour on day 36; oral thioguanine once daily on days 36-49; cytarabine IV continuously on days 38-41 and 45-48; and methotrexate IT on days 38 and 45.
  * Arm II (protocol III x 2 or 3 courses and interim maintenance therapy [IMT]) (SR-2, IR-2, or HR-1): Patients receive dexamethasone orally or IV three times daily on days 1-14 followed by a taper; vincristine sulfate IV and doxorubicin hydrochloride IV over 1 hour on days 1 and 8; and asparaginase IV over 1 hour on days 1, 4, 8, and 11. Patients then receive cyclophosphamide IV over 1 hour on day 15; oral thioguanine once daily on days 15-28; cytarabine IV continuously on days 17-20 and 24-27; and methotrexate IT on days 17 and 21 (and day 1 if there is initial CNS involvement). Approximately 1 week after completion of protocol III (course 1), patients receive IMT for 10 weeks (SR group) or 4 weeks (IR and HR groups) as described below. Approximately 1 week after completion of IMT, patients receive protocol III as above (course 2). Approximately 1 week after completion of protocol III (course 2), patients in IR and HR group receive IMT for another 4 weeks followed by another course of protocol III (course 3) 1 week later.

    * IMT: Patients receive oral methotrexate once weekly and oral mercaptopurine daily.
  * Arm III (HR-2): Patients receive 1 of the following regimens according to local practices:

    * Regimen HR-2A: Patients receive protocol II as in arm I, rest 1 week and receive IMT for 4 weeks. Approximately 1 week later, patients receive another course of protocol II.
    * Regimen HR-2B: Patients receive treatment as in 3-block consolidation regimen with 3 weeks between each block. Approximately 3 weeks later, patients receive protocol II as in arm I.
  * Cranial radiotherapy (CRT) during reinduction: CNS positive patients (CNS status 3) receive CRT after completion of protocol II (SR, IR, HR-2B) or during the first 1.5-2.5 weeks of IMT (SR, IR, HR-2A). SR and IR patients with T-cell ALL and HR patients receive prophylactic CRT at these same time periods.

Beginning 2 weeks after completion of reinduction (some patients in HR group also undergo allogeneic stem cell transplantation, as described below), patients proceed to maintenance therapy.

* Maintenance therapy (MT): Patients receive oral mercaptopurine once daily and methotrexate IV once weekly. Each patient subgroup (except HR patients undergoing transplantation) receives MT for a period that brings the total weeks of treatment to 104 weeks, as follows:

  * SR: Patients receive MT for 74 weeks (SR-1) or 61 weeks (SR-2).
  * IR: Patients receive MT for 74 weeks (IR-1) or 57 weeks (IR-2).
  * HR: Patients receive MT for 58 weeks (HR-1), 62 weeks (HR-2A), or 63 weeks (HR-2B).

Patients with BCP-ALL and in group SR-1 or IR-1 also receive methotrexate IT once in weeks 4, 8, 12, and 16 of MT. Patients with BCP-ALL and in group SR-2 receive methotrexate IT in weeks 4 and 8 of MT.

* Allogeneic stem cell transplantation (ASCT): Some patients in HR group may undergo ASCT (usually bone marrow, but may be peripheral blood or umbilical cord stem cells), (at the time of reinduction therapy) beginning 3-4 weeks after the completion of second protocol III (HR-1), the first protocol II (HR-2A), or completion of the 3-block consolidation regimen (HR-2B).

  * Under 2 years old: Patients receive oral busulfan every 6 hours on days -8 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 1 hour on days -3 and -2, and then undergo ASCT on day 0.
  * At least 2 years old: Patients undergo total body irradiation twice daily on days -6 to -4 and receive etoposide IV over 4 hours on day -3, and then undergo ASCT on day 0. Fractionated local radiotherapy, if required, is administered on days -14 to -7.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically proven acute lymphoblastic leukemia (ALL)
* No relapse of a previously unrecognized ALL
* Patients must meet one of the following risk criteria:

  * Standard-risk (SR) group meeting all of the following criteria:

    * Blasts < 1,000/μL in peripheral blood (PB) on day 8
    * Aged 1 to < 6 years
    * Initial WBC < 20,000/μL
    * M1 (5%) or M2 (≥ 5% to < 25%) blasts in bone marrow on day 15
    * M1 marrow on day 33
  * Intermediate-risk (IR) group meeting all of the following criteria:

    * Aged < 1 or ≥ 6 years and/or WBC ≥ 20,000/μL
    * Blasts < 1,000/μL in PB on day 8
    * M1 or M2 marrow on day 15
    * M3 (≥ 25%) marrow on day 15 OR meets SR criteria but M3 marrow on day 15 and M1 marrow on day 33
  * High-risk (HR) group meeting ≥ 1 of the following criteria:

    * Meets IR criteria and M3 marrow on day 15 (not SR and M3 on day 15)
    * Blasts ≥ 1,000/μL in PB on day 8
    * M2 or M3 marrow on day 33
    * Translocation t(9;22) [BCR/ABL+] (Philadelphia chromosome-positive) or t(4;11) [MLL/AF4+]
* No secondary ALL

PATIENT CHARACTERISTICS:

* No Down syndrome
* No other major disease that prohibits study treatment (e.g., severe congenital heart disease)
* Not requiring significant therapy modification owing to study therapy-associated complications
* No complications due to other interventions
* No one with missing data that are needed for the differential diagnosis, or for selection of the proper therapy arm

PRIOR CONCURRENT THERAPY:

* No steroids or cytostatic drugs within four weeks prior to start of study therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4000 (Estimated)
Dates: Start 2002-11; Primary Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival
Event-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stary, MD, Principal Investigator — University Hospital, Motol
Locations (1):
- University Hospital Motol, Prague, Czechia

REFERENCES:
- [Derived] Zuna J, Moericke A, Arens M, Koehler R, Panzer-Grumayer R, Bartram CR, Fischer S, Fronkova E, Zaliova M, Schrauder A, Stanulla M, Zimmermann M, Trka J, Stary J, Attarbaschi A, Mann G, Schrappe M, Cario G. Implications of delayed bone marrow aspirations at the end of treatment induction for risk stratification and outcome in children with acute lymphoblastic leukaemia. Br J Haematol. 2016 Jun;173(5):742-8. doi: 10.1111/bjh.13989. Epub 2016 Feb 23. PMID 26913693
- [Derived] Stary J, Zimmermann M, Campbell M, Castillo L, Dibar E, Donska S, Gonzalez A, Izraeli S, Janic D, Jazbec J, Konja J, Kaiserova E, Kowalczyk J, Kovacs G, Li CK, Magyarosy E, Popa A, Stark B, Jabali Y, Trka J, Hrusak O, Riehm H, Masera G, Schrappe M. Intensive chemotherapy for childhood acute lymphoblastic leukemia: results of the randomized intercontinental trial ALL IC-BFM 2002. J Clin Oncol. 2014 Jan 20;32(3):174-84. doi: 10.1200/JCO.2013.48.6522. Epub 2013 Dec 16. PMID 24344215